CLINICAL TRIAL: NCT00880529
Title: Does Continuous Subcutaneous Paravertebral Infusion of Bupivicaine With the ON-Q Pain Relief System vs. Standard IV Pain Management Decrease Ventilator Dependence in Trauma Patients With Multiple Rib Fractures
Brief Title: Pain Relief for Ventilated Patients With Multiple Rib Fractures Using the ON-Q Pain Relief System
Acronym: ON-Q
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: low enrollment, 2 pts enrolled no data every analyzed investigator left the institution
Sponsor: The Cooper Health System (Other)
Responsible Party: Principal Investigator, Ashley Shapiro, Principal investigator, The Cooper Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-118
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Rib Fractures
Keywords: rib fractures; ventilator; ON-Q; analgesia
MeSH Terms: conditions — Rib Fractures; Agnosia | interventions — Passive Cutaneous Anaphylaxis; Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ON-Q (Experimental): Subcutaneous bupivicaine administration and IV opioid medication if necessary
  Interventions: Device: ON-Q bupivicaine administration
- IV opioids alone (Active Comparator): Standard therapy with IV opioid administration
  Interventions: Drug: IV opioid administration

INTERVENTIONS:
Device: ON-Q bupivicaine administration — continuous subcutaneous bupivicaine drip
  Other Names: ON-Q, bupivicaine
  Arms: ON-Q
Drug: IV opioid administration — Patient controlled analgesia with IV narcotics
  Other Names: PCA, morphine
  Arms: IV opioids alone

SUMMARY:
The purpose of this study is to find out if patients having the ON-Q post-op Pain Relief System for pain management of multiple rib fractures will require fewer ventilator days, and will need less IV pain medicine to control their pain, and as a result have improved respiratory function during their recovery.

The standard of care for providing pain relief for rib fractures is to use an opioid drug that is injected into the vein but also has side effects. Increased doses can lead to over sedation and consequently lead to difficulty with breathing. The ON-Q pain relief systems uses a local anesthetic under the skin. The anesthetic is called bupivicaine, and it is delivered from a thin tube approximately 10 inches long is tunneled under the skin along the back and parallel to the spine. The medication is stored in an elastic pump which delivers a slow continuous drip of medication from multiple holes in the tubing. Subjects will be randomized to either standard intravenous opioid pain management or the ON-Q pain relief device with supplemental opioid medication if needed. The device will remain in use until the subjects are able to breathe without the ventilator.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* 3 or more rib fractures
* Intubated ready for weaning from ventilator support
* FI02 < 50%
* Peep < 10cm H2O

Exclusion Criteria:

* < 18 years of age
* Pregnant
* Unable to communicate pain status
* Allergy to local anesthetics
* Coagulopathy
* Skin lesions or abnormalities from previous injury or surgery
* < 3 rib fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Time from weaning process initiation to discontinuation of ventilatory support | Time will be measured in hours from initation of ventilator weaning to no ventilatory support needed

SECONDARY OUTCOMES:
total dose of narcotics given will be identified and reported as mcg or mg each 24 hour period that ON-Q pain pump is being used. | each 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia R Fusco, DO, Principal Investigator — The Cooper Health System
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States